CLINICAL TRIAL: NCT02443337
Title: A Phase II Study of the Combination of LY3023414 and Necitumumab After First-Line Chemotherapy for Metastatic Squamous Non-small Cell Carcinoma of the Lung
Brief Title: A Study of LY3023414 and Necitumumab in Squamous Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study stopped due to lack of efficacy.
Sponsor: Eli Lilly and Company (Industry)
Collaborators: SCRI Development Innovations, LLC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15799; I6A-MC-CBBE (Other: Eli Lilly and Company)
Record Dates: First submitted 2015-05-11; First posted 2015-05-13 (Estimated); Results first posted 2020-12-09 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2018-01

CONDITIONS: Non-small Cell Lung Cancer Metastatic
MeSH Terms: interventions — LY3023414; necitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LY3023414 + Necitumumab (Experimental): 200 milligrams (mg) LY3023414 administered orally twice daily and 800 mg necitumumab administered intravenously (IV) on day 1 and day 8 of each cycle (21 day cycles). Participants may continue to receive treatment until discontinuation criteria are met.
  Interventions: Drug: LY3023414; Drug: Necitumumab

INTERVENTIONS:
Drug: LY3023414 — Administered orally
Drug: Necitumumab — Administered IV
  Other Names: LY3012211; IMC-11F8

SUMMARY:
The main purpose of this study is to evaluate the safety and activity of the study drug known as LY3023414 in combination with necitumumab in participants with metastatic squamous non-small cell lung cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed squamous advanced NSCLC (Stage IV).
* Participants must have progressed on one prior line of platinum-based chemotherapy in the advanced or metastatic setting.
* Measurable disease as measured by response evaluation criteria in solid tumors (RECIST) criteria v 1.1.
* Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 or 1.
* Able to swallow the study drugs whole.
* Adequate organ function.
* Women of childbearing potential must have a negative serum or urine pregnancy test performed ≤ 7 days prior to start of treatment. Women of childbearing potential or men with partners of childbearing potential must use effective birth control measures during treatment and during the 3 months following completion of study treatment.

Exclusion Criteria:

* Participants who have received > 1 prior line of chemotherapy in the advanced or metastatic setting. (Immunotherapy will not be considered a line of chemotherapy.)
* Prior treatment with a PI3K/mTOR inhibitor, epidermal growth factor receptor (EGFR) inhibitor, and/or necitumumab.
* History of brain metastases unless irradiated ≥ 2 weeks prior to first study treatment and stable without requirement of corticosteroids.
* Have serious pre-existing medical conditions.
* Have insulin-dependent diabetes mellitus. Participants with a type 2 diabetes mellitus are eligible if adequate control of blood glucose level is obtained by oral anti-diabetics.
* Women who are pregnant or breast-feeding.
* Clinically significant electrolyte imbalance ≥ Grade 2.
* Currently receiving treatment with therapeutic doses of warfarin sodium. Low molecular weight heparin and oral Xa inhibitors are allowed.
* Have initiated treatment with bisphosphonates or approved receptor activator of nuclear factor kappa-B ligand (RANK-L) targeted agents (e.g. denosumab) ≤ 28 days prior to Day 1 of Cycle 1.
* Concurrent serious infection requiring parenteral antibiotic therapy.
* Have a second primary malignancy that in the judgment of the investigator and Medical Monitor may affect the interpretation of results.
* Have an active, known fungal, bacterial, and/or known viral infection.
* History of arterial or venous embolism within 3 months prior to study enrollment. If the embolism occurred >3 and <6 months, the participant is eligible provided appropriate treatment according to institutional standard of care is ensured.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2015-07; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (14):
- United States (14):
  - Southern Cancer Center, P.C., Mobile, Alabama
  - Ironwood Cancer & Research Centers, Chandler, Arizona
  - Comprehensive Cancer Care and Research Institute of Colorado, Englewood, Colorado
  - Florida Cancer Specialists, Fort Myers, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Florida Cancer Specialists, St. Petersburg, Florida
  - Palm Beach Cancer Institute, West Palm Beach, Florida
  - Research Medical Center, Kansas City, Missouri
  - Oncology Hematology Care Inc., Cincinnati, Ohio
  - Chattanooga Oncology Hematology, Chattanooga, Tennessee
  - SMO Sarah Cannon Research Inst., Nashville, Tennessee
  - Tennessee Oncology, Nashville, Tennessee
  - Center for Cancer and Blood Disorders, Fort Worth, Texas
  - University of Virginia Health, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Lilly provides access to the individual patient data from studies on approved medicines and indications as defined by the sponsor specific information on ClinicalStudyDataRequest.com.
  This access is provided in a timely fashion after the primary publication is accepted. Researchers need to have an approved research proposal submitted through ClinicalStudyDataRequest.com. Access to the data will be provided in a secure data sharing environment after signing a data sharing agreement.

REFERENCES:
- See also: Click here for more information about this study: A Study of LY3023414 and Necitumumab in Squamous Lung Cancer — http://www.lillytrialguide.com/EN/studies/cancer/cbbe

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants completed the study if they had objective progressive disease (PD), stable disease (SD), complete response (CR) or partial response (PR).
Groups:
- Lead in Cohort LY3023414 + Necitumumab; Post Lead in Cohort LY3023414 + Necitumumab: 200 milligrams (mg) LY3023414 administered orally twice daily and 800 mg necitumumab administered intravenously (IV) on day 1 and day 8 of each cycle (21 day cycles). Participants may continue to receive treatment until discontinuation criteria are met.
Period: Overall Study
Arm/Group | Lead in Cohort LY3023414 + Necitumumab | Post Lead in Cohort LY3023414 + Necitumumab
Started | 15 | 16
Received at Least One Dose of Study Drug | 15 | 16
Completed | 10 | 14
Not Completed | 5 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Clinical Progressive Disease | 3 | 0
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Lead in Cohort LY3023414 + Necitumumab | Post Lead in Cohort LY3023414 + Necitumumab | Total
Number analyzed (Participants) | 15 | 16 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.0 (10.18) | 68.1 (5.77) | 67.1 (8.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 13 | 11 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 15 | 16 | 31
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 14 | 14 | 28
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 16 | 31

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Complete Response (CR), Partial Response (PR) or Stable Disease (SD) at 6 Months: Disease Control Rate (DCR)
Description: RECIST v 1.1 was used to assess tumor response.The 6-month DCR was defined as the number of participants with PFS > 6 months (or 26 weeks, to accommodate the scheduled tumor assessment at week 24 be delayed by up to 2 weeks) divided by number of participants with baseline tumor assessment.
  Target Lesions:CR was defined as the disappearance of all target lesions. PR was at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.SD was neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD,taking as reference the smallest (nadir) sum of diameters since the treatment started.
  Non-Target Lesions:CR was defined as disappearance of all non-target lesions and normalization of tumor markers.All lymph nodes must be non-pathological in size (<10 millimeters(mm) short axis).SD was defined as the persistence of one or more non-target lesions and/or persistence of tumor marker level above the normal limits.
Time Frame: 6 Months
Population: All participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lead in Cohort LY3023414 + Necitumumab | Post Lead in Cohort LY3023414 + Necitumumab
Number analyzed (Participants) | 15 | 16
percentage of participants | 6.6 [0.2 to 31.9] | 25.0 [7.3 to 52.4]

2. Secondary Outcome: Percentage of Participants Achieving Complete Response (CR) or Partial Response (PR): Objective Response Rate (ORR)
Description: RECIST v 1.1 was used to assess tumor response. ORR for a given participant was based on objective responses determined from data obtained up to: progression, the last evaluable assessment in the absence of progression, or initiation of subsequent anticancer therapy. Participants for whom an objective response cannot be determined or for who the best objective response is not evaluable (NE) were considered non-responders.
  Target Lesions: CR was defined as the disappearance of all target lesions. PR was at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  Non-Target Lesions: CR was defined as disappearance of all non-target lesions and normalization of tumor markers. All lymph nodes must be non-pathological in size (<10 mm short axis). The ORR percentage was calculated as the number of participants with best objective response of CR or PR divided by the number of participants with measurable disease at baseline.
Time Frame: Baseline to Objective Disease Progression or Initiation of Subsequent Anticancer Therapy (Up To 3 Months)
Population: All participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lead in Cohort LY3023414 + Necitumumab | Post Lead in Cohort LY3023414 + Necitumumab
Number analyzed (Participants) | 15 | 16
percentage of participants | 0.00 [0.00 to 21.8] | 0.00 [0.00 to 20.6]

3. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from enrollment until the date of disease progression per RECIST v 1.1 or death by any cause.Participants who had not progressed or died at the time of assessment were censored at the time of the last date of tumor assessment.Participants who are enrolled but do not receive treatment and participants who have no evaluable visits will be censored on day 1.Participants who received new anti-cancer therapy before disease progression or death will be censored to the last tumor assessment date prior to the new anti-cancer therapy.
  Target Lesions:PD is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest(nadir) sum since the treatment started, or the appearance of one or more new lesions. Requires not only 20% increase, but absolute increase of a minimum of 5 mm over sum.
  Non-Target Lesions(NTL):PD is defined as appearance of one or more new lesions and/or unequivocal progression of existing NTL.
Time Frame: Enrollment to Measured Progressive Disease or Death from Any Cause (Up To 12 Months)
Population: All participants who received at least one dose of study drug. Participants censored: Lead in Cohort 1 LY3023414 + Necitumumab= 4 and Post Lead in Cohort LY3023414 + Necitumumab=3
Measure: Median (95% Confidence Interval); unit: Days
Groups:
- Lead in Cohort LY3023414 + Necitumumab; Post Lead in Cohort LY3023414 + Necitumumab: LY3023414 administered orally twice daily and necitumumab administered intravenously (IV) on day 1 and day 8 of each cycle (21 day cycles). Participants may continue to receive treatment until discontinuation criteria are met.
Arm/Group | Lead in Cohort LY3023414 + Necitumumab | Post Lead in Cohort LY3023414 + Necitumumab
Number analyzed (Participants) | 15 | 16
Days | 81 [35 to 168] | 81 [36 to 206]

4. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from enrollment until the date of death by any cause. Participants lost follow up or did not die at the time of assessment were censored at the time of the last known alive date.
Time Frame: Enrollment to Death from Any Cause (Up To 16 Months)
Population: All participants who received at least one dose of study drug. Participants censored: Lead in Cohort 1 LY3023414 + Necitumumab=4 and Post Lead in Cohort LY3023414 + Necitumumab=9
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Lead in Cohort LY3023414 + Necitumumab | Post Lead in Cohort LY3023414 + Necitumumab
Number analyzed (Participants) | 15 | 16
Days | 102 [57 to 285] | 279 [85 to NA] — The study was terminated early and therefore participants were not followed long enough to determine the upper level of the confidence Interval.

5. Secondary Outcome: Pharmacokinetics (PK): Minimum Concentration (Cmin) of LY3023414 and Necitumumab
Description: Minimum Concentration (Cmin) of LY3023414 and Necitumumab
Time Frame: Cycle 1 Day 8, and Cycle 3 Day 8 (pre-dose, end of necitumumab infusion and 1 hour post-necitumumab infusion), Cycle 2 Day 1, Cycle 4 Day 1
Population: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram/milliliter (ng/mL)
Groups:
- LY3023414: 200 milligrams (mg) LY3023414 administered orally twice daily.
- Necitumumab: 800 mg necitumumab administered intravenously (IV) on day 1 and day 8 of each cycle (21 day cycles).
Arm/Group | LY3023414 | Necitumumab
Number analyzed (Participants) | 17 | 26
Nanogram/milliliter (ng/mL)
  Cycle 1 Day 8 | 14 (172) | 69500 (28)
  Cycle 2 day 1: number analyzed (Participants) | 17 | 23
  Cycle 2 day 1 | NA (NA) — LY3023414 samples were below limit of quantification because only predose samples were collected. | 54000 (60)
  Cycle 3 Day8: number analyzed (Participants) | 3 | 5
  Cycle 3 Day8 | 9.73 (221) | 121000 (36)
  Cycle 4 Day 1: number analyzed (Participants) | 17 | 7
  Cycle 4 Day 1 | NA (NA) — LY3023414 samples were below limit of quantification because only predose samples were collected. | 104000 (56)

6. Secondary Outcome: Pharmacokinetics: Maximum Concentration (Cmax) of LY3023414 and Necitumumab
Description: Maximum Concentration (Cmax) of LY3023414 and Necitumumab
Time Frame: Cycle 1 Day 8, and Cycle 3 Day 8 (pre-dose, end of necitumumab infusion and 1 hour post-necitumumab infusion)
Population: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Necitumumab: 800 mg necitumumab administered intravenously (IV) on day 1 and day 8 of each cycle (21 day cycles). Participants may continue to receive treatment until discontinuation criteria are met.
Arm/Group | LY3023414 | Necitumumab
Number analyzed (Participants) | 23 | 26
ng/mL
  Cycle 1 Day 8 | 738 (103) | 318000 (27)
  Cycle 3 Day 8: number analyzed (Participants) | 3 | 6
  Cycle 3 Day 8 | 1302 (70) | 345000 (14)

ADVERSE EVENTS:
Time Frame: Up To 330 Days
Description: All participants who received at least one dose of study drug.
Arm/Group | Lead in Cohort LY3023414 + Necitumumab | Post Lead in Cohort LY3023414 + Necitumumab
All-Cause Mortality (participants affected / at risk) | 11/15 | 6/16
Serious Adverse Events (participants affected / at risk) | 3/15 | 5/16
Other Adverse Events (participants affected / at risk) | 15/15 | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lead in Cohort LY3023414 + Necitumumab (N=15) | Post Lead in Cohort LY3023414 + Necitumumab (N=16)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia fungal (Infections and infestations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lead in Cohort LY3023414 + Necitumumab (N=15) | Post Lead in Cohort LY3023414 + Necitumumab (N=16)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 3 (4)
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 2 (4)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Cyanosis (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Tricuspid valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Deafness (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Cataract (Eye disorders) | 0 (0) | 1 (2)
Dry eye (Eye disorders) | 0 (0) | 1 (1)
Lacrimation increased (Eye disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 2 (3)
Visual impairment (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (3)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 4 (7)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 10 (28)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hyperchlorhydria (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (5) | 11 (19)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Paraesthesia oral (Gastrointestinal disorders) | 1 (2) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (2) | 3 (5)
Vomiting (Gastrointestinal disorders) | 3 (3) | 5 (9)
Asthenia (General disorders) | 2 (2) | 1 (1)
Chills (General disorders) | 2 (2) | 1 (1)
Disease progression (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 7 (8) | 11 (17)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 2 (4) | 3 (9)
Oedema peripheral (General disorders) | 0 (0) | 3 (4)
Pain (General disorders) | 2 (3) | 1 (1)
Pyrexia (General disorders) | 1 (2) | 4 (5)
Temperature intolerance (General disorders) | 0 (0) | 1 (1)
Thirst (General disorders) | 0 (0) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (2)
Herpes zoster (Infections and infestations) | 1 (2) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia fungal (Infections and infestations) | 0 (0) | 1 (1)
Rash pustular (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 3 (3)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase (Investigations) | 1 (3) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase (Investigations) | 1 (5) | 0 (0)
Blood alkaline phosphatase (Investigations) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Blood chloride decreased (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (3)
Blood magnesium decreased (Investigations) | 1 (1) | 1 (1)
Blood phosphorus decreased (Investigations) | 1 (1) | 0 (0)
Electrocardiogram qt prolonged (Investigations) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (8)
Urine ketone body present (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 3 (4) | 4 (6)
Decreased appetite (Metabolism and nutrition disorders) | 5 (5) | 5 (5)
Dehydration (Metabolism and nutrition disorders) | 4 (4) | 4 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (2) | 3 (4)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 4 (6)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2) | 5 (15)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 2 (4)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (2)
Headache (Nervous system disorders) | 3 (4) | 1 (2)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 2 (4)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 3 (4)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 3 (3)
Mental status changes (Psychiatric disorders) | 1 (1) | 1 (1)
Nervousness (Psychiatric disorders) | 0 (0) | 1 (1)
Restlessness (Psychiatric disorders) | 1 (1) | 0 (0)
Chromaturia (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 1 (2)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 2 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 7 (8)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 8 (13) | 4 (5)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (4) | 5 (7)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (4)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (8)
Rash generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (4)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 2 (2)
Hot flush (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 2 (2)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Superior vena cava syndrome (Vascular disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The study stopped due to lack of efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2015-12-16): https://cdn.clinicaltrials.gov/large-docs/37/NCT02443337/Prot_000.pdf
  • Statistical Analysis Plan (2015-12-28): https://cdn.clinicaltrials.gov/large-docs/37/NCT02443337/SAP_001.pdf